CLINICAL TRIAL: NCT02976428
Title: Randomized Controlled Trial of Sensor Guided Knee Balancing Compared to Standard Balancing Technique in Total Knee Arthroplasty
Brief Title: Conventional vs. Sensor Guided Soft Tissue Balancing in TKA RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Mitch Winemaker, Chief Orthopedic Surgery, Hamilton Health Sciences Juravinski Hospital, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HAGRP01
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Total Knee Arthroplasty
Keywords: knee soft tissue balancing; sensor-guided; range of motion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Soft Tissue Balancing (Active Comparator): In the control group where the sensor device is not used in optimization of knee balance and alignment, definitive implants will be cemented in place and the sensor trial inserted using a thickness based on prior standard bearing insert trialing. Peak load data will be captured intraoperatively through full ROM. Custom shims will be affixed to the sensor to replicate thickness of the standard trial. The knee will then be cycled and loads recorded in the medial and lateral compartments at 10, 45 and 90 degrees of flexion. The surgeon will be blinded to the sensor output and the system will be located outside of their visual field.
  Interventions: Procedure: Standard Soft Tissue Balancing
- Sensor Guided Soft Tissue Balancing (Experimental): In the experimental group where the sensor device is used to optimize balance and alignment, the sensor trial will be inserted and tibial baseplate rotated until medial and lateral femoral contact points are parallel on the sensor output. Quantitative balance is defined as a mediolateral intercompartmental loading difference of ≤15 pounds. Flexion balance is achieved when femoral contact point position is within the midposterior third of the tibial insert and intercompartmental loads are balanced. Loads in the medial and lateral compartments are recorded at 10, 45 and 90 degrees. If compartment loads differ by >15 lbs between compartments, unbalanced, further soft tissue release/bone resection will be done to achieve a side to side compartment pressure difference of <15 lbs through ROM.
  Interventions: Procedure: Sensor Guided Soft Tissue Balancing

INTERVENTIONS:
Procedure: Sensor Guided Soft Tissue Balancing — Primary TKR with soft tissue balancing with a sensor guided device.
  Other Names: Triathlon (Stryker, Mahwah, NJ); Verasense (OrthoSensor Inc., Dania Beach, FL)
  Arms: Sensor Guided Soft Tissue Balancing
Procedure: Standard Soft Tissue Balancing — Primary TKR with soft tissue balancing with a standard of care manual tensiometer device.
  Other Names: Triathlon (Stryker, Mahwah, NJ)
  Arms: Standard Soft Tissue Balancing

SUMMARY:
To ensure a successful outcome after total knee replacement (TKR) soft tissue balance and proper implant position are very important during the surgical procedure. Soft tissues are structures in the knee including ligaments, muscles, tendons, and menisci that stabilize and cushion the knee joint. Lack of proper soft tissue balance or imprecise implant positioning may result in knee stiffness, pain, instability and limited range of motion (ROM). This may result in implant failure and the need for revision surgery. As part of standard practice orthopedic surgeons use a manual knee balancer device to help guide soft tissue balancing to achieve optimal knee balance. New sensor-assisted technology can provide surgeons with measurable information to help achieve soft tissue balancing, providing surgeons with immediate visual feedback during the surgery. This feedback, transmitted wirelessly by the sensor, gives surgeons electronic information on soft tissue balance and implant position.The purpose of this study is to determine if a sensor guided soft tissue balancing device (Verasense) is more effective at balancing the knee during surgery as compared to standard soft tissue balancing performed with a manual balancer device.

DETAILED DESCRIPTION:
The study is that of a prospective double-blind randomized controlled trial of patients presenting for elective primary TKR to compare the outcomes of TKR using conventional soft tissue balancing with a tensiometer device versus augmenting the soft tissue balancing with the OrthoSensor VerasenseTM sensor device. The primary outcome will be rate of unbalanced TKRs based on the quantitative Verasense definition of a well balanced knee defined as a mediolateral intercompartmental loading difference of ≤15 pounds through ROM. Secondary outcomes include differences in clinical outcome scores and patient satisfaction among sensor guided cases and controls.

Patients will be randomized to receive TKR with the Triathlon total knee system (Stryker) in the case and control group according to: (1) control group with standard balancing techniques used and sensor data obtained in blinded fashion and not used to balance the TKR implant, (2) experimental case group with sensor guided balancing where sensor data is used to balance the TKR within defined parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective primary unilateral TKR for a diagnosis of osteoarthritis to be performed at the study site by the primary investigators
* Willingness and ability to give informed consent.

Exclusion Criteria:

* Inflammatory arthropathy
* Ligament insufficiencies
* Contraindications to posterior cruciate retaining TKR including: deformity >15 degrees or fixed-flexion contracture >15 degrees
* Previous high tibial osteotomy
* Scheduled to undergo sequential bilateral TKR under one anesthetic
* Scheduled to undergo revision TKR surgery
* Neuromuscular disorder limiting mobility or ability to comply with physiotherapy
* Previous recurrent deep knee infection
* Major bone loss requiring structural bone graft or augmented components
* Functionally limiting peripheral vascular disease
* Patients receiving associated worker's compensation benefits (WSIB)
* Ethanol/drug abuse/psychiatric disorder
* Inability or unwillingness to give written informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Rate of Unbalanced TKRs | Intraoperative at end of procedure prior to wound closure
  The rate of unbalanced TKRs will be assessed based on the Verasense sensor device quantitative definition of a well balanced knee. A well balanced knee is defined as having a mediolateral intercompartmental loading difference of ≤15 pounds through ROM [Gustke et al., Walker et al].

SECONDARY OUTCOMES:
Knee Society Score | Preoperative, 6 weeks, 6 months and 1 year postoperative
  Overall clinical function as measured by Knee Society Score
Oxford Knee Score | Preoperative, 6 weeks, 6 months and 1 year postoperative
  Subjective function as measured by Oxford Knee Score patient report outcome measure
Patient satisfaction | 1 year postoperative
  Patient satisfaction with total knee replacement; likert scale
Clinical knee function: varus/valgus alignment | Preoperative, intraoperative, 6 weeks, 6 months and 1 year postoperative
  Assessment of clinical knee function
Clinical knee function: anteroposterior stability | Preoperative, intraoperative, 6 weeks, 6 months and 1 year postoperative
  Assessment of clinical knee function
Clinical knee function: extension lag | Preoperative, intraoperative, 6 weeks, 6 months and 1 year postoperative
  Assessment of clinical knee function
Clinical knee function: anatomic alignment | Preoperative, intraoperative, 6 weeks, 6 months and 1 year postoperative
  Assessment of clinical knee function
Clinical knee function: knee ROM | Preoperative, intraoperative, 6 weeks, 6 months and 1 year postoperative
  Assessment of clinical knee function

CONTACTS AND LOCATIONS:
Overall Officials: Mitch Winemaker, MD, FRCSC, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences Juravinski Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gustke KA, Golladay GJ, Roche MW, Elson LC, Anderson CR. A new method for defining balance: promising short-term clinical outcomes of sensor-guided TKA. J Arthroplasty. 2014 May;29(5):955-60. doi: 10.1016/j.arth.2013.10.020. Epub 2013 Oct 24. PMID 24269069
- [Background] Walker PS, Meere PA, Bell CP. Effects of surgical variables in balancing of total knee replacements using an instrumented tibial trial. Knee. 2014 Jan;21(1):156-61. doi: 10.1016/j.knee.2013.09.002. Epub 2013 Sep 19. PMID 24103411